CLINICAL TRIAL: NCT06785064
Title: OPT-X: OPTimizing an EXtended Care Intervention to Promote Weight Loss Maintenance
Brief Title: Optimizing an Extended Care Intervention to Promote Weight Loss Maintenance
Acronym: OPT-X
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Gareth R. Dutton PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300013598; R01DK139059 (NIH)
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Obesity Prevention; Weight Change; Weight Loss; Weight Loss Maintenance
Keywords: weight loss maintenance; weight loss; weight change; health behavior; reduced food variety; ACT workshop; buddy support; home-based resistance training; weight training
MeSH Terms: conditions — Body Weight Changes; Weight Loss; Health Behavior | interventions — Resistance Training; Palliative Care

STUDY DESIGN:
Intervention Model Description: Investigators used the multiphase optimization strategy (MOST) as the ideal approach for the proposed study as, with the four proposed intervention components, identifying an optimal intervention through a single randomized controlled trial (RCT) with multiple arms or through multiple RCTs would be methodologically inefficient and resource-intensive. Given this, investigators rely on the eloquent and rigorous MOST-based optimization design, which leverages factorial experimentation to identify an optimal set of intervention component(s). In a factorial experiment, the goal is not to compare individual experimental conditions (in this case, 16 conditions), but to use combinations of conditions to estimate the main and interaction effects of the intervention components. Thus, numerous intervention components can be evaluated simultaneously while utilizing the entire randomized sample.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Package 1: No WLM Components (No Intervention): Participants will receive education and support for weight loss maintenance only.
- Package 2: One WLM Component - BTS (Active Comparator): Participants will receive education and support for weight loss maintenance and Buddy Training and Support.
  Interventions: Behavioral: Buddy Training and Support (BTS)
- Package 3: One WLM Component - HBRT (Active Comparator): Participants will receive education and support for weight loss maintenance and Home-based Resistance Training
  Interventions: Behavioral: Home-based Resistance Training (HBRT)
- Package 4: Two WLM Components - HBRT+BTS (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Home-based Resistance Training and Buddy Training and Support.
  Interventions: Behavioral: Home-based Resistance Training (HBRT); Behavioral: Buddy Training and Support (BTS)
- Package 5: One WLM Component - ACT (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Acceptance and Commitment (ACT) Workshops.
  Interventions: Behavioral: Acceptance and Commitment (ACT) Workshops
- Package 6: Two WLM Components - BTS+ACT (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Buddy Training and Support and ACT Workshops.
  Interventions: Behavioral: Buddy Training and Support (BTS); Behavioral: Acceptance and Commitment (ACT) Workshops
- Package 7: Two WLM Components - HBRT+ACT (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Home-based Resistance Training and ACT Workshops.
  Interventions: Behavioral: Home-based Resistance Training (HBRT); Behavioral: Acceptance and Commitment (ACT) Workshops
- Package 8: Three WLM Components - HBRT+BTS+ACT (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Home-based Resistance Training, Buddy Training and Support, and ACT Workshops.
  Interventions: Behavioral: Home-based Resistance Training (HBRT); Behavioral: Buddy Training and Support (BTS); Behavioral: Acceptance and Commitment (ACT) Workshops
- Package 9: One WLM Component - RFV (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Reduced Food Variety.
  Interventions: Behavioral: Reduced Food Variety (RFV)
- Package 10: Two WLM Components - RFV+BTS (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Reduced Food Variety and Buddy Training and Support
  Interventions: Behavioral: Reduced Food Variety (RFV); Behavioral: Buddy Training and Support (BTS)
- Package 11: Two WLM Components - RFV+HBRT (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Reduced Food Variety and Home-based Resistance Training.
  Interventions: Behavioral: Reduced Food Variety (RFV); Behavioral: Home-based Resistance Training (HBRT)
- Package 12: Three WLM Components - RFV+HBRT+BTS (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Reduced Food Variety, Home-based Resistance Training, and Buddy Training and Support.
  Interventions: Behavioral: Reduced Food Variety (RFV); Behavioral: Home-based Resistance Training (HBRT); Behavioral: Buddy Training and Support (BTS)
- Package 13: Two WLM Components - RFV+ACT (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Reduced Food Variety and ACT Workshops.
  Interventions: Behavioral: Reduced Food Variety (RFV); Behavioral: Acceptance and Commitment (ACT) Workshops
- Package 14: Three WLM Components - RFV+BTS+ACT (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Reduced Food Variety, Buddy Training and Support, and ACT Workshops.
  Interventions: Behavioral: Reduced Food Variety (RFV); Behavioral: Buddy Training and Support (BTS); Behavioral: Acceptance and Commitment (ACT) Workshops
- Package 15: Three WLM Components - RFV+HBRT+ACT (Active Comparator): Participants will receive education and support for weight loss maintenance as well as Reduced Food Variety, Home-based Resistance Training, and ACT Workshops.
  Interventions: Behavioral: Reduced Food Variety (RFV); Behavioral: Home-based Resistance Training (HBRT); Behavioral: Acceptance and Commitment (ACT) Workshops
- Package 16: Four WLM Components: RFV+HBRT+BTS+ACT (Experimental): Participants will receive education and support for weight loss maintenance as well as Reduced Food Variety, Home-based Resistance Training, Buddy Training and Support, and ACT Workshops.
  Interventions: Behavioral: Reduced Food Variety (RFV); Behavioral: Home-based Resistance Training (HBRT); Behavioral: Buddy Training and Support (BTS); Behavioral: Acceptance and Commitment (ACT) Workshops

INTERVENTIONS:
Behavioral: Reduced Food Variety (RFV) — Participants engaged in reduced food variety (RFV) will be asked to choose a few high-calorie, low nutrient main meals and snacks to eat regularly. At the beginning of each month, they will choose one main meal (entrée) to eat at least 2 times a week and one snack food to eat at least 4 times a week within the month. They will have the option to keep or change their main meal and snack options from month to month.
  Arms: Package 10: Two WLM Components - RFV+BTS; Package 11: Two WLM Components - RFV+HBRT; Package 12: Three WLM Components - RFV+HBRT+BTS; Package 13: Two WLM Components - RFV+ACT; Package 14: Three WLM Components - RFV+BTS+ACT; Package 15: Three WLM Components - RFV+HBRT+ACT; Package 16: Four WLM Components: RFV+HBRT+BTS+ACT; Package 9: One WLM Component - RFV
Behavioral: Home-based Resistance Training (HBRT) — Participants assigned to receive home-based resistance training (also called strength training or lifting weights) will be asked to engage in at-home exercises that strengthen muscles at least 2 days each week (≤45 minutes per home session) and track their progress. They will be asked to attend 6, 1-hour group-based skills training workshops (in-person and/or remotely via Zoom) during the first two months of Phase 2 to learn these skills. They will receive exercise plans and equipment (sets of dumbbells, a rack to hold the dumbbells, and an exercise mat) needed to complete exercises.
  Other Names: Strength Training; Resistance Training; Weight Lifting; Lifting Weights
  Arms: Package 11: Two WLM Components - RFV+HBRT; Package 12: Three WLM Components - RFV+HBRT+BTS; Package 15: Three WLM Components - RFV+HBRT+ACT; Package 16: Four WLM Components: RFV+HBRT+BTS+ACT; Package 3: One WLM Component - HBRT; Package 4: Two WLM Components - HBRT+BTS; Package 7: Two WLM Components - HBRT+ACT; Package 8: Three WLM Components - HBRT+BTS+ACT
Behavioral: Buddy Training and Support (BTS) — Participants assigned to buddy training and support will be asked to identify an eligible friend or family member who is over 18 years old that can be their "buddy". Study staff will contact the buddy to be sure they are eligible, willing, and have all the details they need. The participant's buddy will be asked to attend up to 6 training sessions with the study staff, so they can learn the best ways to support the participant during the program. After the buddy completes training, they will be asked to check in with the participant 1-2 times each week about their progress.
  Other Names: Buddy Support
  Arms: Package 10: Two WLM Components - RFV+BTS; Package 12: Three WLM Components - RFV+HBRT+BTS; Package 14: Three WLM Components - RFV+BTS+ACT; Package 16: Four WLM Components: RFV+HBRT+BTS+ACT; Package 2: One WLM Component - BTS; Package 4: Two WLM Components - HBRT+BTS; Package 6: Two WLM Components - BTS+ACT; Package 8: Three WLM Components - HBRT+BTS+ACT
Behavioral: Acceptance and Commitment (ACT) Workshops — Participants assigned to receive Acceptance and Commitment (ACT) Workshops will be asked to attend 6, 1-hour group-based skills training workshops (in-person and/or remotely via Zoom) during the first three months of Phase 2. These workshops will help them develop skills to handle tough thoughts about weight control, keep their values in mind, and be mindful of their decisions and the impact of their decisions related to weight control. They will also be asked to apply ACT skills regularly during the rest of Phase 2.
  Other Names: ACT Workshop
  Arms: Package 13: Two WLM Components - RFV+ACT; Package 14: Three WLM Components - RFV+BTS+ACT; Package 15: Three WLM Components - RFV+HBRT+ACT; Package 16: Four WLM Components: RFV+HBRT+BTS+ACT; Package 5: One WLM Component - ACT; Package 6: Two WLM Components - BTS+ACT; Package 7: Two WLM Components - HBRT+ACT; Package 8: Three WLM Components - HBRT+BTS+ACT

SUMMARY:
The purpose of this study is to find out what combination of components, if any, offers the best support for keeping weight off after someone loses weight. Long term weight loss maintenance is a challenge for many people who lose weight. There are many strategies, or components, people may use to avoid regain, but investigators do not know if there is a best, or optimal, combination of such components that can be done without adding a lot of cost or other burdens for people.

* The primary goal of this clinical trial is to identify the optimal package that maximizes weight loss maintenance.
* The study also wants to understand the reasons why these components may work and if certain components help specific sub-groups of people.

Participants will engage in a 16-week Phase 1 Weight Loss Program. Participants who lose 5% or more of their weight during that program will continue to Phase 2 Extended Care and be randomly assigned to 0, 1, 2, 3, or all of four methods of weight loss maintenance. They will use their assigned package for 12 months. Researchers will compare 16 different possible combinations of components and learn which of the 16 packages offers the best support for keeping weight off.

The four components participants could be assigned to in Phase 2 are:

1. Reduced Food Variety: Limiting the variety of foods participants eat by having them choose a few high-calorie, low nutrient foods to eat regularly
2. Home-based Resistance Training: Engaging in exercises that build strength from the comfort of the participant's own home
3. Buddy Training and Support: Having a friend or "buddy" get trained to support the participant
4. Acceptance and Commitment (ACT) Workshops: Having participants learn skills to handle tough thoughts and feelings about weight control in a healthy way

Participants will have their weight measured and complete surveys 4 times if they complete both Phase 1 and Phase 2. During Phase 1, participants will attend weekly group sessions and be in touch with a study staff member investigators call a Wellness Coach. During Phase 2, participants will stay in touch with their Wellness Coach, use their assigned package, and answer questions about their experience periodically.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Body mass index (BMI) >30 kg/m2
* Has regular access to internet (to access Zoom videoconferencing platform)
* If indicated during screening, willing to obtain medical clearance for exercise from their healthcare provider prior to enrollment

Exclusion Criteria:

* Current or recent (past 6 months) use of prescription weight loss medications
* Weight loss >10 pounds in past 6 months (other than postpartum)
* Pregnancy or anticipating pregnancy
* Another household member already participating in the study
* Participation in another randomized research project
* Uncontrolled hypertension (blood pressure >160/100 mm Hg at screening)
* Any of the following other medical conditions: myocardial infarction or cerebrovascular accident within the last 6 months; unstable angina within the past 6 months; NYHA Class III or IV congestive heart failure; type 1 diabetes; and chronic lung diseases that limit physical activity
* Unable to identify potential buddy (i.e., adult friend or family member) for extended care intervention phase
* Residing >50 miles from the university (to attend assessment visits)
* Planning to relocate out of the area in the next 18 months
* Does not have internet access
* Unwilling or unable to do any of the following: give informed consent; read/understand English; accept random assignment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in weight from time of randomization to 12 months | 12 months
  The primary outcome of the study is the change in weight measurement from the time of randomization (after Phase 1 initial weight loss/the beginning of Phase 2) until the follow up visit 12 months later. Participants' body weight will be measured to the nearest 0.1 kg at each point using a calibrated electronic scale. The change between these two measures will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States